CLINICAL TRIAL: NCT04184986
Title: The Czech National Fabry Disease Screening Study in Patients Diagnosed With Non-infectious Inflammatory Bowel Disease, Functional Dyspepsia or Irritable Bowel Syndrome
Brief Title: Screening of Fabry Disease in Patients With GI Symptoms
Acronym: GiFD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: General University Hospital, Prague (Other)
Collaborators: Charles University, Czech Republic (Other); Klinické centrum ISCARE (Unknown); Amicus Therapeutics (Industry)
Responsible Party: Principal Investigator, Gabriela Dostálová, Principal Investigator, General University Hospital, Prague
Other Study IDs: 1
Record Dates: First submitted 2019-12-01; First posted 2019-12-04 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Fabry Disease
Keywords: Fabry Disease, gastrointestinal, GI symptoms, screening
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — dry blood test
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- inflammatory bowel disease: 100-150 pts with dg. inflammatory bowel disease
  Interventions: Diagnostic Test: dry blood test
- unspecific GI symptoms: 100-150 pts unspecific GI symptoms
  Interventions: Diagnostic Test: dry blood test

INTERVENTIONS:
Diagnostic Test: dry blood test — screening test for Fabry disease

SUMMARY:
Fabry disease screening study in patients diagnosed with gastrointestinal tract (GIT) disease, i.e. with the diagnosis of non-infectious inflammatory bowel disease, functional dyspepsia or irritable bowel syndrome in particular, is a project designed as a pilot study of Centre for Fabry disease, General University Hospital in Prague, and Clinical Centre ISCARE Prague, focused on improving the diagnosis and care of patients with Fabry disease in the Czech Republic.

Fabry disease, (FD) is an X-linked inherited, rare, progressive disorder of glycosphingolipid metabolism affecting multiple organs resulting in organ dysfunction. The earlier diagnosis is made the earlier treatment is started the better outcome patients have.

There are screening programs in cardiology, nephrology, neurology or ophtalmology fields. But not only cardiovascular, renal or eye symptoms are present. Very common are also GI symptoms in Fabry disease patient population. This is the first screening of FAbry disease in GI symptom patients.

DETAILED DESCRIPTION:
Fabry disease screening study in patients diagnosed with gastrointestinal tract (GIT) disease, i.e. with the diagnosis of non-infectious inflammatory bowel disease, functional dyspepsia or irritable bowel syndrome in particular, is a project designed as a pilot study of Centre for Fabry disease, General University Hospital in Prague, and Clinical Centre ISCARE Prague, focused on improving the diagnosis and care of patients with Fabry disease in the Czech Republic.

Introduction Fabry (Anderson-Fabry) disease is a progressive multiorgan X-linked lysosomal storage disease. The disease is caused by a deficiency of the enzyme alpha-galactosidase A. The enzymatic defect leads to accumulation of enzyme substrate in various tissue types. The affected tissue types include the vascular endothelium of several organs involving kidneys, heart, nervous system, and GIT. Glycolipids accumulation triggers function impairment of affected organs and their subsequent failure. The disease is X-linked and most female heterozygotes develop milder symptoms or the disease manifests later in life than in affected hemizygous man. The disease burden is milder in women due to second X-chromosome.

A typical clinical picture can emerge in males as early as childhood. The onset of clinically evident symptoms manifests with attacks of neuropathic pain of the extremities, followed with early manifestation of hypohidrosis and development of skin lesions - angiokeratomata. In affected hemizygous males, sign of renal damage can be detected even in the second decade, representing already considerable renal damage leading to ultimate organ failure with the need for hemodialysis or kidney transplantation. The first gastrointestinal symptoms occur. From the third decade onwards, both males and females can present neurological symptoms such as white matter lesions as well as stroke, mostly of ischemic nature. Cardiac involvement is characterized by a thickening of the ventricular wall occurring in the third decade in men and approximately ten years later in women. The finding may remind of classical sarcomeric hypertrophic cardiomyopathy in its full extent, including left ventricular outflow tract obstruction. Patients suffer dyspnea, arrhythmias and chest pain. In some patients, other classical symptoms and manifestations of Fabry disease may be completely absent, and the patients with predominant or exclusive cardiac involvement are sometimes referred to as having a cardiac variant.

Most patients with Fabry disease report GI symptoms of diarrhea, with frequent abdominal pain attacks and increased flatulence. Defecation frequency varies, most often 4-6 times a day, which patients consider normal. However, more than 8-times-a-day evacuation episodes are common. Unlike in inflammatory bowel diseases such as Crohn's or ulcerative colitis, no blood or mucus in stool is present. Some patients, on the other hand, complain of severe constipation. Patients with Fabry disease may then be followed-up under diagnosis of non-infectious inflammatory bowel disease, functional dyspepsia or irritable bowel syndrome.

The diagnosis of Fabry disease is based on the evaluation of the defect enzyme activity level in plasma or leukocytes in males. In females, this test is less effective as the enzyme activity levels can reach near normal levels. Thus, sequencing of DNA of the GLA gene is necessary for a diagnosis in most females. they are diagnosed by DNA analysis for a mutation responsible for enzyme deficiency. In women Prior to sequencing, level of the lyso-Gb3 biomarker can be tested and the finding of elevated lyso-Gb3 should be the ultimate requirement for genetic testing.

Treatment is based on enzyme replacement therapy. Two approved treatments are available in Europe. Chaperones, small molecules that stabilize defective α-galactosidase A enzyme, and allow its residual activity to be increased, have recently been introduced.

Aim of the Study The aim of the study is to screen patients for Fabry disease in medical centers concentrating patients diagnosed idiopathic inflammatory bowel disease to better determine the prevalence of this disease in the Czech Republic.

Methods This is the first screening study organized by of Centre for Fabry disease in cooperation with departments of gastroenterology. The Clinical Centre ISCARE Prague is invited to participate. The aim of the Study is to obtain samples of dry blood spot along with a elementary medical history of the gastrointestinal tract disease from a study population of 500-800 patients at least that were diagnosed with idiopathic inflammatory bowel disease, functional dyspepsia or irritable bowel syndrome. The study has been evaluated and is approved by the Multicenter Ethics Committee of the General University Hospital in Prague (EC General University Hospital in Prague).

Patients of both sexes older than 18 years and under 60 years of age are enrolled in the Study. Other inclusion criteria include previous examination and follow-up for the GIT symptoms, usually the above-mentioned diagnoses.

During a routine outpatient follow-up, samples of 4 drops of blood will be drawn from the patient finger as per the instructions. Alternatively, the blood sample will be taken during another routine blood test. Enzyme activity evaluation and/or genetic tests will be carried out by the ARCHIMED Lie Science Laboratories GmbH (Austria). The dry blood spot kits will first be sent to Center for Fabry Disease at II. Internal Clinic of Cardiology and Angiology of the First Faculty of Medicine and General University Hospital, where they will be anonymized and sent for processing. At the same time, the attending physician will complete a brief questionnaire on the patient's basic clinical data (age, gender, GIT symptoms, other symptoms of Fabry disease). Patients with a positive test result will then be invited to the Center for Fabry Disease at the General University Hospital in Prague, where specific treatment will be considered in accordance with the current criteria for covering by the health insurance company. Patients do not receive any financial compensation for their participation in the study. Patients invited to the Center for Fabry Disease will be reimbursed for their travel expenses.

The project is a pilot study. If patients suffering Fabry disease are identified, a nationwide screening will follow.

ELIGIBILITY:
Inclusion Criteria:

* 18 -60years old males, females
* ICF sign
* GI symptoms and/or inflammatory bowel disease

Exclusion Criteria:

* do not agree with dry blod test or genetic testing

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: GI symptaomatic patients seen by gastroenetologists for their GI symptoms
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
prevalence of Fabry disease in GI symptomatic patients | 1 year
  To assess prevalence of Fabry disease in GI symptomatic participants, alpha-galactosidase enzymatic activity will be determined in samples of dry blood spot of patients with some medical history of idiopathic inflammatory bowel disease, functional dyspepsia or irritable bowel syndrom in a study population of 500-800 patients.

CONTACTS AND LOCATIONS:
Overall Officials: gabriela Dostálová, MD, PhD., Study Director — General University Hospital, Prague; Ales Linhart, prof., MD., Principal Investigator — General University Hospital, Prague
Locations (1):
- General Teaching Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
after first 6 months first data available - number of screened/positive/negative pts
Supporting Information: Study Protocol
Time Frame: 2 years
Access Criteria: email ask